CLINICAL TRIAL: NCT05378490
Title: The Akershus Study of Ischemic Stroke and Thrombolysis -1 (ASIST-1) Epidemiology, Clinical and Radiological Presentation and Treatment of Cerebrovascular Disease and Stroke Mimics in a Norwegian Population
Brief Title: The Akershus Study of Ischemic Stroke and Thrombolysis -1
Acronym: ASIST-1
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Collaborators: University of Oslo (Other); Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Espen Saxhaug Kristoffersen, Associate professor, MD, PhD, University Hospital, Akershus
Other Study IDs: ASIST-1
Record Dates: First submitted 2022-01-19; First posted 2022-05-18 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Stroke, Acute; Intracerebral Hemorrhage; Stroke, Ischemic; TIA
MeSH Terms: conditions — Stroke; Cerebral Hemorrhage; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Intravenous thrombolysis (IVT): All patients treated with IVT in the acute stroke care pathway 2012-2025
- Intracerebral hemorrhage (ICH): All patients with intracerebral hemorrhage 2012-2019
- Acute ischemic stroke (AIS) and Intracerebral hemorrhage (ICH): All patients with acute ischemic stroke or intracerebral hemorrhage 2015-2017
- Stoke care pathway: All patients admitted to the stroke care pathway (ischemic stroke, intracerebral hemorrhage, transient ischemic attack and stroke mimics) 2015-2017
- Endovascular treatment: All stroke patients treated with endovascular treatment 2012-2025
- Cerebellar hematoma (cICH): All patients with cerebellar hematoma 2008-2019

SUMMARY:
This observational study comprises consecutively patients with cerebrovascular diseases admitted to the Stroke Unit at Akershus University Hospital in Norway. Akershus University Hospital is the largest emergency care hospital in Norway and has a catchment area covering a population of 550.000, which is approximately 10 % of the Norwegian population and reasonably representative according to data from Statistics Norway. The hospital is public and serving both as a primary hospital and a university hospital. Due to the Norwegian, national, all-covering health-insurance, all patients enter the hospital and are considered for further in-patient care on the same conditions. The hospital has a stroke unit classified as a comprehensive stroke center according to European Stroke Organisation standards. Acute stroke management follows national and international guidelines. Overall, the ASIST-1 study will investigate management, outcome and prognosis of stroke and stroke care pathways and later follow up in primary care using several approaches combining existing clinical data from a representative population with different Norwegian health registries. Parts of the study are retrospective with prospective follow-up by health registries and parts of the study are prospective.

DETAILED DESCRIPTION:
Aims

i) to describe the use of the stroke fast track and the proportion of all those evaluated in the fast track actually treated with intravenous thrombolysis, ii) to identify reasons for not giving thrombolysis in patients with acute stroke symptoms < 4.5 hours at admission to hospital, iii) to investigate whether or not some of these patients that did not receive thrombolysis actually could have been given thrombolysis, iv) to investigate the outcome of patients in the stroke fast track treated or not treated with thrombolysis (or endovascular thrombectomy), v) to investigate differences between stroke and stroke mimics for patients reaching the hospital within or outside the thrombolysis time window of 4.5 hours, vi) to investigate differences between stroke subtypes (both ischemic and hemorrhagic) and stroke mimics for patients reaching the hospital within or outside the thrombolysis time window of 4.5 hours, vii) to investigate outcomes for patients with acute ischemic stroke, hemorrhagic stroke, transient ischemic attack (TIA) or stroke mimics, viii) to investigate predictors and factors related to functional outcome for patients with acute ischemic stroke, hemorrhagic stroke, TIA or stroke mimics, ix) to describe the epidemiology of large vessel occlusions in a representative hospital population, x) to describe hemorrhagic stroke in a representative hospital population, xi) whether risk factors, acute blood pressure variability or imaging (CT, angiography, perfusion or MRI) may predict diagnosis or outcome at discharge, 3 months, 12 months and 2 years for the ASIST-1 population, xii) whether risk factors, acute blood pressure variability or imaging (CT, angiography, perfusion or MRI) may predict outcome at discharge, 3 months, 12 months and 2 years for different sub-types of stroke, xiii) to investigate readmission until 5 years after initial admission for acute stroke symptoms xiv) whether deep learning-based assessment of acute phase CT, CT perfusion and CT angiography can reliably identify infarct core, penumbra and large-vessel occlusion, estimate reliably collateral score, predict risk of adverse events, or guide target blood pressure during acute and subacute ischemic stroke specialized treatment, xv) whether deep learning-based assessment of acute phase CT, CT perfusion and CT angiography or MRI can predict clinical outcome in different types of stroke, xvi) whether deep learning-based assessment of acute phase CT, CT perfusion, CT angiography or MRI can be used for automatic detection of hematoma volume and localization in hemorrhagic stroke xvii) whether deep learning-based assessment of acute phase CT or MRI can predict risk of new incidents after a hemorrhagic stroke and thus guide the clinicians to whether or not patients should be started/re-started on anti-platelet therapy or anticoagulation xviii) to investigate secondary prevention after different subtypes of stroke and the adherence of statins, anti-platelet therapy, anti-coagulation and blood pressure treatment up to 5 years after stroke, also in relation to readmission rates and long-term mortality xix) to prospectively investigate quality in terms of treatment, complications, prognosis and predictive factors of all patients given thrombolysis and/or thrombectomy at Ahus 2019-2025 xx) to investigate the changes in prehospital delay, the use of stroke fast track, stroke pathways and treatment over time (2012-2025).

ELIGIBILITY:
Inclusion Criteria:

* Cerebrovascular diseases (acute ischemic stroke, intracerebral hemorrhage, transient ischemic attack) or stroke mimics

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. IVT treated patients 2012-2025 (2012-2018 retrospective, 2019-2025 prospective)
  2. All patients with ICH (2011-2019 retrospective, 2020-2025 prospective)
  3. All patients with acute ischemic stroke or ICH (2015-2018 retrospective, 2019-2025 prospective)
  4. All patients admitted to the stroke care pathway (stroke/mimics 2015-2017)
  5. All stroke patients treated with endovascular treatment 2012-2025 (2012-2018 retrospective, 2019-2025 prospective)
  6. All patients with cerebellar hematoma 2008-2022 (retrospective)
  Data will be linked with data from general practitioners, Municipal Patient Registry (KRP/KUHR), Norwegian Patient Registry (NPR), Norwegian Prescription Database (NorPD), Norwegian Stroke registry, Cause of Death Registry (DÅR)
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Large vessel occlusion in a representative Norwegian population | Baseline 2015-2017
  Incidence of large vessel occlusion 2015-2017
Functional status | 3 months
  modified Rankin Scale (mRS) 0-6 (0 normal, 6 dead) for all groups
Functional status | Index discharge from hospital, usually up to 1 month
  modified Rankin Scale (mRS) 0-6 (0 normal, 6 dead) for all groups
Mortality | In-hospital, usually up to 1 month
  Number dead vs total number of cases all groups
Mortality | 3 months
  Number dead vs total number of cases all groups
Mortality | 12 months
  Number dead vs total number of cases all groups
Mortality | 24 months
  Number dead vs total number of cases all groups
Mortality | 5 years
  Number dead vs total number of cases all groups
Diagnostic precision of different published clinical screening scales of stroke and large vessel occlusion | Baseline 2015-2017
  Diagnostic precision, accuracy and validity of clinical screening scales

SECONDARY OUTCOMES:
Reasons for not giving thrombolysis in patients with acute stroke symptoms < 4.5 hours | Baseline 2015-2017
  Number of cases treated with thrombolysis vs number of cases evaluated in the acute stroke care pathway
Functional outcome of patients in the stroke fast track treated or not treated with thrombolysis (or endovascular thrombectomy), | 3 months
  Modified Rankin Scale (mRS) 0-6 (0 normal, 6 dead)
Mortality of patients in the stroke fast track treated or not treated with thrombolysis (or endovascular thrombectomy), | 3 months
  Mortality
Functional outcome after 1 year of patients in the stroke fast track treated or not treated with thrombolysis (or endovascular thrombectomy), | 1 year
  modified Rankin Scale (mRS) 0-6 (0 normal, 6 dead)
Mortality after 1 year of patients in the stroke fast track treated or not treated with thrombolysis (or endovascular thrombectomy), | 1 year
  Mortality
Functional outcome at discharge of patients in the stroke fast track treated or not treated with thrombolysis (or endovascular thrombectomy), | Discharge after index admission, usually up to 1 month
  modified Rankin Scale (mRS) 0-6 (0 normal, 6 dead)
Mortality at discharge of patients in the stroke fast track treated or not treated with thrombolysis (or endovascular thrombectomy), | Discharge after index admission, usually up to 1 month
  Mortality
Re-admission | Baseline to five years
  Number of new re-admission among included patients
New prescriptions | Baseline to five years
  Type of new prescriptions
Use of anti-coagulation in the long-term | Baseline to five years
  Number of patients treated with anti-coagulation
Use of anti-platelet therapy in the long-term | Baseline to five years
  Number of patients treated with anti-platelet therapy
Use of cholesterol-lowering drugs in the long-term | Baseline to five years
  Number of patients treated with cholesterol-lowering drugs
Use of anti-hypertensive drugs in the long-term | Baseline to five years
  Number of patients treated with anti-hypertensive drugs
Use of anti-diabetics in the long-term | Baseline to five years
  Number of patients treated with anti-diabetics
Health care utilisation | Baseline to five years
  Number of new health care system contacts
Prehospital delay | 2012-2025
  Changes in prehospital delay (minutes)
Time of stroke fast track | 2012-2025
  Changes in the use of stroke fast track (minutes)
Use of stroke fast track | 2012-2025
  Changes in the use of stroke pathways (proportion)
Treated in the stroke fast track | 2012-2025
  Changes in proportion treated over time
Blood pressure variability baseline (diastolic, systolic and pulse pressure) | Baseline
  Different BP measurements from general practitioners, ambulance, hospital and follow-up
Blood pressure variability discharge after index (diastolic, systolic and pulse pressure) | Discharge after index admission, usually up to 1 month
  Different BP measurements from general practitioners, ambulance, hospital and follow-up
Blood pressure variability follow-up (diastolic, systolic and pulse pressure) | Follow-up (3 to 6 months)
  Different BP measurements from general practitioners, ambulance, hospital and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Espen S. Kristoffersen, MD, PhD, Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lørenskog, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Could be possible, but must be approved by Medical Ethics Committee in Norway

REFERENCES:
- [Background] Bergh E, Jahr SH, Ronning OM, Askim T, Thommessen B, Kristoffersen ES. Reasons and predictors of non-thrombolysis in patients with acute ischemic stroke admitted within 4.5 h. Acta Neurol Scand. 2022 Jul;146(1):61-69. doi: 10.1111/ane.13622. Epub 2022 Apr 21. PMID 35445395
- [Background] Larsen KT, Selseth MN, Jahr SH, Hillestad V, Koubaa N, Sandset EC, Ronning OM, Kristoffersen ES. Prehospital Blood Pressure and Clinical and Radiological Outcomes in Acute Spontaneous Intracerebral Hemorrhage. Stroke. 2022 Dec;53(12):3633-3641. doi: 10.1161/STROKEAHA.121.038524. Epub 2022 Oct 17. PMID 36252098
- [Background] Larsen KT, Sandset EC, Selseth MN, Jahr SH, Koubaa N, Hillestad V, Kristoffersen ES, Ronning OM. Antithrombotic Treatment, Prehospital Blood Pressure, and Outcomes in Spontaneous Intracerebral Hemorrhage. J Am Heart Assoc. 2023 Mar 7;12(5):e028336. doi: 10.1161/JAHA.122.028336. Epub 2023 Mar 4. PMID 36870965
- [Background] Meinel TR, Wilson D, Gensicke H, Scheitz JF, Ringleb P, Goganau I, Kaesmacher J, Bae HJ, Kim DY, Kermer P, Suzuki K, Kimura K, Macha K, Koga M, Wada S, Altersberger V, Salerno A, Palanikumar L, Zini A, Forlivesi S, Kellert L, Wischmann J, Kristoffersen ES, Beharry J, Barber PA, Hong JB, Cereda C, Schlemm E, Yakushiji Y, Poli S, Leker R, Romoli M, Zedde M, Curtze S, Ikenberg B, Uphaus T, Giannandrea D, Portela PC, Veltkamp R, Ranta A, Arnold M, Fischer U, Cha JK, Wu TY, Purrucker JC, Seiffge DJ; International DOAC-IVT, TRISP, and CRCS-K-NIH Collaboration; DOAC-IVT Writing Group; Kagi G, Engelter S, Nolte CH, Kallmunzer B, Michel P, Kleinig TJ, Fink J, Ronning OM, Campbell B, Nederkoorn PJ, Thomalla G, Kunieda T, Poli K, Bejot Y, Soo Y, Garcia-Esperon C, Ntaios G, Cordonnier C, Marto JP, Bigliardi G, Lun F, Choi PMC, Steiner T, Ustrell X, Werring D, Wegener S, Pezzini A, Du H, Marti-Fabregas J, Canovas-Verge D, Strbian D, Padjen V, Yaghi S, Stretz C, Kim JT. Intravenous Thrombolysis in Patients With Ischemic Stroke and Recent Ingestion of Direct Oral Anticoagulants. JAMA Neurol. 2023 Mar 1;80(3):233-243. doi: 10.1001/jamaneurol.2022.4782. PMID 36807495
- [Background] MacIntosh BJ, Liu Q, Schellhorn T, Beyer MK, Groote IR, Morberg PC, Poulin JM, Selseth MN, Bakke RC, Naqvi A, Hillal A, Ullberg T, Wasselius J, Ronning OM, Selnes P, Kristoffersen ES, Emblem KE, Skogen K, Sandset EC, Bjornerud A. Radiological features of brain hemorrhage through automated segmentation from computed tomography in stroke and traumatic brain injury. Front Neurol. 2023 Sep 28;14:1244672. doi: 10.3389/fneur.2023.1244672. eCollection 2023. PMID 37840934